CLINICAL TRIAL: NCT04020172
Title: Can Dobutamine and Goal-Directed Fluid Therapy Improve Tissue Oxygenation in Deep Inferior Epigastric Perforator (DIEP) Flap Breast Reconstruction Surgery? Randomized Controlled Trial
Brief Title: Improving Tissue Oxygenation in Breast Reconstruction Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Glenio Mizubuti (MD, PhD) (Other)
Responsible Party: Sponsor-Investigator, Dr. Glenio Mizubuti (MD, PhD), Dr. Glenio Mizubuti (MD, MSc, FRCPC), Anesthesiologist, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ANAE-341-19
Record Dates: First submitted 2019-07-08; First posted 2019-07-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Perioperative Tissue Oxygenation
Keywords: tissue flap oxygenation; DIEP flap breast reconstruction surgery
MeSH Terms: interventions — Dobutamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dobutamine + Goal-Directed Fluid Therapy (Experimental): All patients will receive a baseline infusion of Ringer's lactate at 2 ml/kg/h to satisfy maintenance fluid requirements. The intervention will commence at anesthesia induction and continue for up to 4 hours postoperatively. In addition to maintenance fluids, patients will receive 250 ml fluid challenges with crystalloid as required until they are no longer fluid responsive. The absence of fluid responsiveness will be defined as the absence of a sustained rise in stroke volume index of at least 10% for 20 minutes or more, at which point, the patient will be considered fluid optimized. At this point, a low-dose dobutamine infusion at a fixed rate (2.5 μg/kg/min) will be commenced and maintained until 4 hours postoperatively. The infusion rate will be halved and/or discontinued if the patient develops tachycardia (heart rate ≥ 100 bpm) for more than 30 minutes despite adequate anesthesia/analgesia and fluid status.
  Interventions: Drug: Dobutamine
- Standard of care (No Intervention): Patients in the control group will also receive a baseline infusion of Ringer's lactate at 2 ml/kg/h to satisfy maintenance fluid requirements, which will be commenced upon admission to the operating room. The anesthetic management will otherwise be according to standard practice. No specific cardiac output monitoring device will be used to guide fluid therapy. Likewise, perioperative dobutamine will not be used unless clinically indicated to improve cardiac function.

INTERVENTIONS:
Drug: Dobutamine — intraoperative fluid administration will be guided by cardiac output monitoring
  Other Names: intraoperative fluid administration
  Arms: Dobutamine + Goal-Directed Fluid Therapy

SUMMARY:
Breast reconstruction is an integral part of breast cancer care. There are two main types of breast reconstruction: alloplastic (using implants), and autologous (using patient's tissue). The latter creates a more natural breast mound, and avoids long-term concerns requiring surgical re-intervention associated with implant-based surgery. The deep inferior epigastric perforator (DIEP) flap is the gold standard technique in autologous breast reconstruction. Complications, however, do occur with DIEP flap surgery and often stem from poor flap perfusion/oxygenation. Hence, the development of strategies to enhance flap perfusion (e.g., optimal perioperative fluid therapy) is essential. Current perioperative fluid therapy is usually guided by subjective criteria which leads to wide variations in fluids administered. We will randomly assign DIEP flap patients to receive optimal (cardiac output-guided) fluid therapy in combination with dobutamine (a medication which has potential to improve flap oxygenation) versus the current standard of care. Flap oxygenation will be monitored via near-infrared spectroscopy in all patients for up to 48 hours postoperatively. Optimal fluid therapy in combination with dobutamine may improve flap oxygenation and thereby, reduce complications.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the effects of perioperative hemodynamic therapy (guided by cardiac output monitoring) on tissue oxygenation during (and after) DIEP flap breast reconstruction surgery. We hypothesize that a low-dose, perioperative dobutamine infusion combined with goal-directed fluid therapy guided by cardiac output monitoring will improve flap perfusion (and, thus, oxygenation) in patients undergoing DIEP surgery.

The primary outcome is tissue oxygenation, measured via near-infrared spectroscopy (NIRS), 45 minutes following vascular re-anastomosis of the DIEP flap within the perfusion zone that is furthest away from the perforator vessels. This zone is the most vulnerable surgical area to ischemia and, therefore, the most likely to reflect the potential benefits of the proposed intervention. In the case of bilateral DIEP flaps, the most vulnerable zone will be assessed in both the left and right breasts.

Secondary outcomes include: (1) tissue oxygenation at baseline (preoperatively), intra-operatively, 1, 2, 4, 8 hours postoperatively, as well as the morning of postoperative days 1 and 2; (2) the amount of intravenous fluids (crystalloids, colloids, blood products) and vasopressors (e.g., phenylephrine, ephedrine, norepinephrine, etc.) administered intraoperatively and up to 4 hours postoperatively; (3) the need for intraoperative surgical vascular re-intervention (i.e., re-anastomosis); (4) laboratory measures including perioperative pH, serum lactate, and hemoglobin measures; (5) the incidence of postoperative nausea and vomiting (PONV); (6) hospital length of stay; (7) any postoperative complications including infection, hematoma and those resulting from flap mal-perfusion (i.e., partial/total flap loss and/or fat necrosis); (8) the need for postoperative intervention for flap-related issues; (9) overall patient satisfaction; and (10) days alive and out of hospital (DAOH) all up until 30 days postoperatively.

Study Design and Duration:

This is a prospective, randomized controlled trial. Forty participants will be randomized to one of two groups (n=20/group) using computer-generated randomization. Patient randomization will be concealed in envelopes and opened only by research staff (not otherwise involved with data collection) and/or the attending anesthesiologist prior to anesthesia induction. Blinding will be maintained until study completion (n=20/group) and verification that all outcome data has been successfully collected for all study participants. Each participant will be monitored perioperatively until postoperative day 2 (or until discharge from hospital) and will receive a 30 day follow-up telephone call.

Patient Population:

Eligible consenting patients scheduled to undergo an elective unilateral or bilateral DIEP flap breast reconstruction surgery under the care of Dr. Martou and/or Dr. Edmunds at the Kingston General Hospital site of Kingston Health Sciences Centre.

Intervention Group:

The intervention will commence from the induction of general anesthesia and continue until 4 hours after surgery. Ringer's lactate (2 ml/kg/h) will be commenced upon admission to the operating room to satisfy maintenance fluid requirements. Cardiac output (CO) and stroke volume index (SVI) will be measured by one of two CO monitors: (1) FloTrac system, Edwards Lifesciences Corporation, Irvine, CA, USA, which attaches to the arterial line already in place in this surgical population; or (2) Starling SV system, Cheetah Medical, Vancouver, WA, USA, a non-invasive CO monitor that utilizes 4 stickers placed on the patient's trunk. No more than 500 ml of intravenous fluid will be administered at anesthesia induction. In addition to the maintenance fluid described previously, patients will receive 250 ml fluid challenges with crystalloid as required until they are no longer fluid responsive. Albumin 5% will also be allowed for fluid challenges at the discretion of the attending anesthesiologist. The absence of fluid responsiveness will be defined as the absence of a sustained rise in SVI of at least 10% for 20 minutes or more, at which point the patient will be considered fluid optimized. At this point, a low-dose dobutamine infusion at a fixed rate (2.5 μg/kg/min) will be commenced and maintained until 4h postoperatively. The infusion rate will be halved and/or discontinued if the patient develops tachycardia (heart rate ≥ 100 bpm) for more than 30 minutes despite adequate anesthesia/analgesia and fluid status (based on the above mentioned intervention). Further fluid challenges will be performed by the attending anesthesiologist with the aim to maintain a maximal value of SVI throughout the case. Postoperatively, the patient will remain in the post-anesthetic care unit (PACU) for a minimum of 4 hours (as per current standard of care) at the end of which, the CO monitoring and the dobutamine infusion will be discontinued, and the patient transferred to a level 2 step-down critical care unit. Ringer's lactate at 2 ml/kg/h will be infused to satisfy maintenance fluid requirements until oral fluid intake is permitted by the surgical team, at which point the maintenance infusion will be stopped. Data collection and follow-up for such patients will be performed as per standard of care.

Control group:

Patients in the control group will also receive a baseline infusion of Ringer's lactate at 2 ml/kg/h to satisfy maintenance fluid requirements, which will be commenced upon admission to the operating room. The anesthetic management will otherwise be according to standard practice. This will include 250 ml fluid challenges with a crystalloid administered at the discretion of the attending anesthesiologist, which is generally guided by pulse rate, arterial pressure, urine output, and/or core-peripheral temperature gradient. Albumin 5% will also be allowed for fluid challenges at the discretion of the attending anesthesiologist. No specific CO monitoring device will be used to guide fluid therapy; however, a CO monitor will be present in the operating room throughout the case to ensure adequate blinding of the surgical team and the research staff with regards to which group the patient had been randomized. Perioperative dobutamine will not be used unless clinically indicated to improve cardiac function. It will not be used as described in this protocol (i.e., intervention group) as it is not currently part of our standard practice in these surgeries; and there is not yet documented evidence to support its use in all DIEP flap patients. We expect that this study addresses this gap and provides evidence as to whether there is benefit to indicate using it routinely. Postoperative care will be similar to the intervention group (except for the CO monitoring and dobutamine infusion in PACU).

A tissue oximeter device (SnapshotNIR, KENT Imaging, Calgary, Canada) will be used for all patients. This is a portable non-invasive monitor that measures tissue oxygen saturation using near-infrared spectroscopy (NIRS) technology with the capability of saving images to allow for subsequent analyses. Measurements are taken by holding the monitor at a standardized (30-cm) distance from the skin area where the oxygen levels are to be measured. Upon admission to the operating room, pre-operative, baseline measurements (with patients breathing ambient air without supplemental oxygen) will be recorded over the abdominal flap tissue, followed by recordings immediately post-induction, 1 hour post-induction, when the abdominal flap is free (and still being perfused by the perforator arteries), prior to clamp removal post-arterial re-anastomosis, and 45 minutes following re-anastomosis. All research personnel dedicated to this study will receive pre-study training regarding perfusion zones and the study outcomes to ensure that oxygenation measures are consistently taken from the same surgical region in relation to the perfusion zones throughout each case. In addition, the surgical team, led by Drs. Martou and Edmunds, will also assist with guiding the intraoperative oxygenation measurements. The surgical team and attending anesthesiologist will be blinded to the KENT oxygenation measurements throughout the perioperative period, and surgery will be guided as per standard of care. The surgical team will also be blinded to group allocation. The ischemic period during which the flap is transferred (reflected by a fall in the oxygen saturation of the flap) as well as the time of flap revascularization (characterized by increased oxygen saturation) will be recorded. Upon completion of the surgical procedure, another NIRS-based monitor (Somanetics INVOS 5100C Cerebral/Somatic Oximeter, Medtronic, Minneapolis, USA) may be applied to the freshly reconstructed graft at the surgeon's discretion. If deemed appropriate, a sticker will be applied over the flap for continuous monitoring of the graft oxygenation for up to 48 hours postoperatively. However, if the surgeon requires the entirety of the graft to be exposed for visual monitoring (as per standard care), a sensor will not be applied and postoperative measures will be recorded at 1, 2, 4, and 8 hours postoperatively, as well as on the morning of postoperative days 1 and 2 using the KENT device. All measures will be consistently taken at the same location. Note that intraoperative oximetry continuous monitoring with the Somanetics INVOS Oximeter is not possible as the sensors cannot be sterilized.

All surgical procedures will be performed by one of two surgeons to minimize variability in patient selection and surgical technique, both predictors of clinical outcomes in microsurgery. Elective DIEP flap surgical procedures and anesthetic management will all be completed in accordance with the standard of care. Perioperative management will be identical in both groups, apart from the hemodynamic monitoring for guiding intravenous fluid therapy, and interventions as described below. In the operating room, the ambient temperature will be set at 20°C and standard monitors will be applied. Invasive monitoring in the form of an arterial line will be established as per current practice. General anesthesia will be induced with propofol and fentanyl followed by rocuronium to facilitate endotracheal intubation; and maintained with sevoflurane (Etsevo=1.5-3.0%) and additional doses of fentanyl and/or hydromorphone administered at the discretion of the attending anesthesiologist. Extra doses of rocuronium will be administered throughout the case for muscle relaxation. A mean arterial pressure (MAP) ≥65 mmHg (or within 20% of baseline) will be targeted throughout the perioperative period. Likewise, all patients will receive standard measures to maintain oxygenation (SpO2 ≥95%), end-tidal CO2 (EtCO2) between 35-40 mmHg, hemoglobin (>8 g/dl), and heart rate (<100 bpm). A warming device (enFlow IV Fluid/Blood Warming System, GE Healthcare, Boston, MA, USA) will be used for intravenous fluids, as well as a forced-air patient warming system (3M Bair Hugger Normothermia System, 3M, St. Paul, MN, USA) in order to maintain normothermia (core temperature 36-37.5°C). Arterial blood gasses will be checked every 2 hours (or more often at the discretion of the attending anesthesiologist) to specifically monitor the pH, SpO2, PaO2, PaCO2, base excess, hemoglobin, and lactate levels as surrogates for tissue perfusion perioperatively. Urine output will be recorded hourly. The total amount of vasopressor, perioperative fluid (crystalloids and Albumin 5%) and blood products, if any, will be recorded. In addition, the following demographic and surgical characteristics will be included: age, body mass index, preoperative hemoglobin and hematocrit, levels, American Society of Anesthesiologists classification, Charlson Comorbidity Index, and total surgical and anesthetic time. Prophylactic intravenous dexamethasone 4 mg on induction of general anesthesia, and ondansetron 4 mg 15 minutes prior to completion of the surgical procedure will be given for prevention of nausea and vomiting. All patients will be managed postoperatively in a high dependency unit (level 2 critical care) and will be given an intravenous patient-controlled analgesia (IV-PCA) with hydromorphone (or an alternative in the case of adverse reactions) for post-operative pain management as per current standard of care. The postoperative goals (up to 48h postoperative) will be similar to the intraoperative period, namely: MAP ≥65 mmHg (or within 20% of baseline), SpO2 ≥95%, PaCO2 35-45 mmHg, hemoglobin >8 g/dl, core temperature between 36-37.5°C, and heart rate <100 bpm. Patients will be contacted and/or their medical record accessed 30 days after surgery to determine whether the patient experiences postoperative complications and/or required medical attention (as per the informed consent). If the patient is successfully contacted, they will be asked about their overall satisfaction.

Rescue Medication & Risk Management:

All anesthesia and surgical procedures are according to standard of care except for the low-dose dobutamine infusion intraoperatively and potentially up to 4 hours postoperatively, the use of CO monitoring to guide fluid administration intraoperatively and up to 4 hours postoperatively, and non-invasive measurements of tissue oxygenation until 48 hours postoperatively. Patients will be intensively monitored and medications will be administered as considered medically necessary (conversely, no medications deemed medically necessary will be withheld as a result of study participation). The main potential side-effect associated with dobutamine is tachycardia. In order to mitigate this risk, our protocol proposes a very low-dose infusion. In addition, the dobutamine infusion rate will be halved and/or discontinued if the patient develops tachycardia (heart rate ≥ 100bpm) for more than 30 minutes despite adequate anesthesia/analgesia and fluid status. In addition, all patients will be intensively monitored while in hospital for any adverse events/complications all of which will be carefully considered in terms of whether they are related to the study intervention or otherwise and action will be taken accordingly.

Premature Withdrawal / Discontinuation Criteria:

One of the limitations of a dobutamine infusion is tachycardia. The infusion rate will be halved and/or discontinued if a patient develops tachycardia (heart rate ≥100 bpm) for more than 30 minutes despite adequate anesthesia/analgesia and fluid status (based on the above mentioned intervention). If the reduced dose does not correct the tachycardia, then the infusion will be turned off. In addition, if at any point attending staff raises concerns about the patient being at an increased risk because of study participation, the intervention will be stopped and the patient removed from the investigation. Also, if at any point (prior to publication), the patient decides they want to withdraw their consent, they will be excluded from the study and none of the information collected from them will be used for research purposes. The study intervention only applies during surgery and potentially for 4 hours after. All study participants will be in a fully monitored setting for the duration of study intervention and beyond for up to 48 hours postoperatively. They will have immediate access to any additional care or intervention if required. Adverse events and serious adverse events (SAE) will be monitored and documented. Study staff will mandatorily report all SAE's and serious unexpected adverse drug reactions (SUSARs) to the investigator for evaluation as soon as they become aware of it. All adverse events will be immediately reported to the Queen's University Health Sciences and Affiliated Teaching Hospitals Research Ethics Board and to the Health Canada, Therapeutic Products Directorate.

If patients are withdrawn from the study, we will continue to enroll patients consecutively until we have met our stipulated sample size of 20 patients per group. For patients who are withdrawn, we will seek permission to retain any data collected (especially demographic information) for comparison of those who were versus were not withdrawn to determine whether they differ in any respect (e.g. are older, etc.). However, if at any point the patient decides they want to withdraw their consent (even afterwards), they will be excluded from the study and none of the information collected from them will be used for study purposes.

Efficacy Variables and Analysis:

Our primary objective is to establish whether the use of minimally invasive CO monitoring for guidance of intravenous fluid administration, combined with low-dose dobutamine infusion (via a treatment algorithm), will increase tissue oxygenation in patients undergoing DIEP flap surgery, measured by near-infrared spectroscopy (NIRS). The primary outcome is tissue oxygenation, measured via NIRS, 45 minutes following vascular re-anastomosis of the DIEP flap within the perfusion zone that is furthest away from the perforator vessels. This zone is the most vulnerable surgical area to ischemia and, therefore, the more likely to reflect the potential benefits of the proposed intervention.

Tissue oxygenation will also be measured at baseline (preoperatively), intraoperatively, 1, 2, 4, 8 hours postoperatively, as well as the morning of postoperative days 1 and 2.

Safety Variables and Analysis:

Invasive monitoring in the form of an arterial line will be established in all patients for intensive monitoring (hemodynamics, etc.), as per standard perioperative care for this surgical procedure. In addition, CO monitoring will be used to guide intravenous fluid administration in the intervention group. Other safety variables collected will include postoperative complications resulting from flap mal-perfusion (i.e., partial/total flap loss and/or fat necrosis); (2) the need for surgical re-intervention for flap-related issues; (3) the amount of intravenous fluids (crystalloids, colloids, blood products) administered intraoperatively; (4) incidence of postoperative nausea and vomiting, infection, and hematoma; (5) hospital length of stay; and (6) days alive and out of hospital (DAOH). Differences in perioperative pH, lactate and hemoglobin levels will also be compared between groups.

Statistical Analysis:

Data will be entered into REDCAP (version 10.6.12) and upon study completion, will be exported to IBM SPSS (version 28.0 for Windows, Armonk, New York 2021) for statistical analysis. Descriptive analyses, including means, standard deviations, medians and quartiles for continuous data, and frequencies and percentages for categorical data, will be completed for all demographic and surgical characteristics, and study outcomes. The underlying distributions of all continuous data will be assessed for normality using the Shapiro Wilk test. Tissue oxygenation will be compared using independent samples t-tests if the data are normally distributed, or the Mann-Whitney U in the event that they are not. Secondary outcomes will be compared between the two groups using the Fisher's Exact or Pearson chi-square tests (as appropriate depending on cell sizes) for categorical data, and independent samples t-tests (or the Mann-Whitney U depending on the underlying distribution) for continuous data. Repeated measures ANOVA, with group as a factor, will be used to compare the tissue oxygenation over time (baseline, 1, 2, 4 and 8 hours post-operatively; as well as baseline, post-operative day 1 and day 2 data). A p-value of <0.05 will be used as the criterion for statistical significance and no adjustment will be made for multiple comparisons. The possibility of a type I error will be acknowledged and the actual p-values will be presented for all comparisons.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' (ASA) Physical Classification I-III;
* Undergoing elective unilateral or bilateral DIEP flap surgery;
* Competent to provide informed consent.

Exclusion Criteria:

* Dementia or neurological impairment;
* Scheduled for DIEP flap combined with any other secondary surgical procedure;
* Documented left ventricular dysfunction (ejection fraction < 40%);
* Contraindication to low-dose dobutamine;
* Body mass index < 18 or > 40 kg/m2;
* Pregnant or lactating;
* Renal insufficiency (eGFR < 30 ml/min/1.73m2);
* Known liver insufficiency (i.e., documented cirrhosis, coagulopathy and/or encephalopathy of hepatic origin).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — No it is not based upon gender identity. However this study is based upon sex because it examines an intervention used during DIEP flap breast reconstruction surgery which is most often performed on women.
Enrollment: 40 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Tissue Flap Oxygenation | 45 min following vascular re-anastomosis
  Tissue oxygenation of the breast flap tissue (measured via near-infrared spectroscopy, NIRS), 45 minutes following vascular re-anastomosis of the DIEP flap within the perfusion zone that is furthest away from the perforator vessels.

SECONDARY OUTCOMES:
Tissue Flap Oxygenation | Immediately preoperatively until up to 48 hours postoperatively
  Tissue oxygenation of the breast flap tissue (measured via near-infrared spectroscopy, NIRS)
Complications Associated with Flap Mal-Perfusion | Immediately postoperatively until 30 days postoperatively
  Partial or total flap loss, necrosis, need for surgical reintervention, etc.
Other Complications | Immediately postoperatively up until 30 days postoperatively
  Incidence of nausea & vomiting, infection, hematoma
Intravenous Fluids | Immediately preoperatively until up to 48 hours postoperatively
  Cumulative amount (of each) of colloids, crystalloids, blood products, vasopressors
Hospital Length of Stay | From date and time of end of surgery until the date and time of discharge from hospital or up to 30 days postoperatively (whichever comes first).
  Length of time from end of surgery to hospital discharge or readiness to discharge (hours)
Patient Satisfaction | Immediately postoperatively until 30 days postoperatively
  Overall patient-reported satisfaction with surgical procedure (scale of 0-10)
DAOH | From date and time of discharge from hospital to 30 days postoperatively
  Days alive and out of hospital

CONTACTS AND LOCATIONS:
Overall Officials: Glenio B. Mizubuti, MD, MSc, FRCPC, Principal Investigator — Queen's University - Anesthesiology
Locations (2):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mizubuti GB, Ho AM, Phelan R, DuMerton D, Shelley J, Vowotor E, Xiong J, Smethurst B, McMullen M, Hopman WM, Martou G, Edmunds RW, Tanzola R. Dobutamine and Goal-Directed Fluid Therapy for Improving Tissue Oxygenation in Deep Inferior Epigastric Perforator (DIEP) Flap Breast Reconstruction Surgery: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Nov 22;12:e48576. doi: 10.2196/48576. PMID 37991835